CLINICAL TRIAL: NCT00381251
Title: An Open-Label, Single-Dose, Randomized, 3-Period, Crossover, Bioequivalence Study Between Two New Formulations of 0.45 mg/1.5 mg Premarin / Medroxyprogesterone Acetate (MPA) Compared With a Reference Formulation of 0.45mg/1.5mg Premarin / MPA (Prempro™) in Healthy Postmenopausal Women.
Brief Title: Study Comparing Bioequivalence of Two New Formulations of Premarin/MPA With Premarin/MPA Reference Formulation.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0713E1-134
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2007-06-11 (Estimated); Status verified 2007-06

CONDITIONS: Postmenopausal Osteoporosis; Postmenopause
Keywords: vaginal atrophy; postmenopausal osteoporosis; menopause; hot flashes
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Hot Flashes

INTERVENTIONS:
Drug: Formulations A and B of Premarin/MPA 0.45 mg/0.5 mg and PREMPRO0.45 mg/0.5 mg

SUMMARY:
This study will compare the bioequivalence of two new investigational combination formulations of Premarin and medroxyprogesterone acetate (MPA) with a currently marketed formulation of Premarin and medroxyprogesterone, Prempro™.

Prempro is indicated for use after menopause in women with a uterus to reduce moderate to severe hot flashes; to treat moderate to severe dryness, itching, and burning, in and around the vagina; and to help reduce your chances of getting osteoporosis (thin weak bones). The purpose of this study is to determine if these new formulations of Premarin and MPA provide the same levels of estrogen and MPA in the blood as Prempro in healthy postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, postmenopausal women ages 35 to 70 years, inclusive.
* Naturally postmenopausal women must not have had a menstrual period for at least six months, but less than 12 months, as confirmed by a blood test; or for at least 12 months with no blood hormone test confirmation. Naturally postmenopausal women must not have had a menstrual period since the age of 54. Surgically menopausal women must have undergone bilateral oophorectomy (removal of both ovaries) at least 5 months prior to the start of the study, and the surgical report may be requested to confirm the surgery date and that the surgery was not due to a cancerous condition.
* Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2006-09; Study Completion 2007-01

PRIMARY OUTCOMES:
Pharmacokinetic blood samples for unconjugated and total (unconjugated plus conjugated) estrogens and MPA will be obtained. The following pharmacokinetic parameters will be determined: Cmax, Tmax, t½, AUC0-T, AUC0-¥.

CONTACTS AND LOCATIONS:
Overall Officials: Trial Manager, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer